CLINICAL TRIAL: NCT01487915
Title: Gemcitabine-Carboplatin Versus Gemcitabine-Oxaliplatin in Cisplatin Un-fit Advanced Urothelial Carcinoma: Randomized Phase II Study
Brief Title: Gemcitabine-Carboplatin Versus Gemcitabine-Oxaliplatin in Cisplatin-unfit Urothelial Carcinoma
Acronym: COACH
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, JLee, Associate professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UOSG-AMC-1001; KCSG-GU10-16 (Other: Korean Cancer Study Group)
Record Dates: First submitted 2011-12-05; First posted 2011-12-08 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Advanced Urothelial Carcinoma
Keywords: Cisplatin-unfit condition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GCb (Active Comparator): Gemcitabine plus Carboplatin
  Interventions: Drug: GCb
- GemOx (Experimental): Gemcitabine plus Oxaliplatin
  Interventions: Drug: GemOx

INTERVENTIONS:
Drug: GCb — Gemcitabine 1000 mg/㎡ D1, D8 plus Carboplatin AUC=4.5 D1 every 3 weeks
  Arms: GCb
Drug: GemOx — Gemcitabine 1000 mg/㎡ D1 plus Oxaliplatin 100 mg/㎡ D1 every 2 weeks
  Arms: GemOx

SUMMARY:
Cisplatin-based chemotherapy is the standard regimen for advanced urothelial carcinoma.

But cisplatin-unfit patients account for up to 30-40% of patients in clinical practice.

Recently reported phase II/III trial of EORTC 30986 comparing gemcitabine/carboplatin (GCb) with MCAVI (Methotrexate, Carboplatin, Vinblastine) suggested that GCb be the preferred regimen over MCAVI based on the response rates, adverse events, and severe acute toxicities.

But the grade 3 or worse toxicities associated with GCb are not infrequent and need more effective and more tolerable regimens.

GemOx has been reported to be effective and have very favorable toxicity profiles.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically of histologically confirmed urothelial carcinoma
* Locally advanced or metastatic disease
* Measurable disease according to RECIST v.1.1
* ECOG PS 0-2
* Cisplatin-unfit condition (any of the followings: NYHA functional class 3, creatinine clearance 30-60 ml/min, and ECOG PS=2)
* Adequate organ function
* Chemotherapy-naive

Exclusion Criteria:

* Histology other than urothelial carcinoma, but squamous cell carcinoma or adenocarcinoma mixed with urothelial carcinoma are allowed
* CNS metastases
* Peripheral neuropathy grade 2 or worse
* Serious medical or surgical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-10; Primary Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Response rate | 12 weeks
  Response rate based on RECIST 1.1

SECONDARY OUTCOMES:
Safety | 12 months
  Safety according to NCI CTCAE v.4.03
Progression-free survival | 1 year
Overall survival | 1 year

CONTACTS AND LOCATIONS:
Locations (5):
- South Korea (5):
  - Keimyeong University Dongsan Medical Center, Daegu
  - Chungnam University Hospital, Daejeon
  - Korea University Anam Hospital, Seoul
  - Asan Medical Center, Seoul
  - Chung Ang University Hospital, Seoul

REFERENCES:
- [Derived] Park I, Kim BS, Lim HY, Kim HJ, Lee HJ, Choi YJ, Park KH, Lee KH, Yoon S, Hong B, Hong JH, Ahn H, Lee JL. Gemcitabine plus carboplatin versus gemcitabine plus oxaliplatin in cisplatin-unfit patients with advanced urothelial carcinoma: a randomised phase II study (COACH, KCSG GU10-16). Eur J Cancer. 2020 Mar;127:183-190. doi: 10.1016/j.ejca.2019.08.034. Epub 2019 Oct 24. PMID 31668839